CLINICAL TRIAL: NCT05227105
Title: Increasing Physical Activity in Rural Pennsylvanians: The PA Moves Trial
Brief Title: PA Moves Trial - Patient Participants
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Kathryn Schmitz, Professor, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: STUDY22110037; R01CA268017 (NIH)
Record Dates: First submitted 2022-01-27; First posted 2022-02-07 (Actual); Last update posted 2025-05-07 (Actual); Status verified 2025-05

CONDITIONS: Overweight or Obesity; Diabetes Mellitus, Type 2; Physical Inactivity
MeSH Terms: conditions — Overweight; Obesity; Diabetes Mellitus, Type 2; Sedentary Behavior | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Physical Activity intervention (Active Comparator): Five physical activity coaching calls with MoveLine and weekly physical activity. Objective tracking of activity with an accelerometer will occur at baseline, after 12 months, and after 24 months.
  Interventions: Behavioral: Physical Activity
- Delayed intervention (Placebo Comparator): Objective tracking of activity with an accelerometer will occur at baseline, after 12 months, and after 24 months.
  Interventions: Behavioral: Delayed intervention

INTERVENTIONS:
Behavioral: Physical Activity — Physical activity will be encouraged up to an amount of 150 minutes per week.
  Arms: Physical Activity intervention
Behavioral: Delayed intervention — Physical activity will be encouraged at the end of the trial.
  Arms: Delayed intervention

SUMMARY:
The purpose of this study is to address physical inactivity in rural populations in Pennsylvania.

DETAILED DESCRIPTION:
People living in rural areas are diagnosed and die from cancer at higher rate than people living in cities. Physical activity has been shown to decrease the risk and occurrence of a variety of cancers, including bladder, breast, colon, endometrial, gastric, kidney, and prostate cancers. Being inactive can cause over 10% of breast and colon cancer cases.

Compared to people living in cities, people living in rural areas tend to be less physically active. They're also more likely to be overweight/obese or have diabetes. Adults who are overweight, obese, or diabetic often have changes in the way their bodies deal with insulin, glucose metabolism, and inflammation. Physical activity is thought to reduce the risk of cancer by improving these issues over time.

Primary care providers and their staff can identify a patient's need for more physical activity, but may not have the time or resources to give advice or assistance. We have set up a telephone-based physical activity coaching program, called the MoveLine, to give inactive patients advice and assistance in becoming more physically active.

The purpose of this study is to determine if referring inactive patients to the MoveLine will help them to be more physically active over time. Approximately 880 people will take part in this research in rural areas of Pennsylvania.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 - 75 at the time of enrollment
* Either overweight/obese (Body Mass Index (BMI) ≥ 25) or diabetic (hemoglobin A1c ≥ 5.7%)
* Physically inactive (defined as < 90 min/week of self-reported structured physical activity)
* Able to speak, read, and understand the English language
* Resides in a rural area of Pennsylvania with a Rural Urban Continuum Code (RUCC) 4 - 9 or Rural-Urban Commuting Area (RUCA) code 4 - 10
* Must be able to provide and understand informed consent
* Primary care patient of one of the participating providers
* Self-report ability to walk ¼ mile
* Access to a telephone

Exclusion Criteria:

* Cardiac exclusion criteria: Class II, III, or IV heart failure as defined by the New York Heart Association (NYHA) functional classification system, history of acute coronary syndromes, uncertain or uncontrolled arrhythmia, uncontrolled hypertension, syncope, acute myocarditis, acute pericarditis, acute endocarditis, acute pulmonary embolus or pulmonary infarction, thrombosis of lower extremities, suspected dissecting aneurysm, pulmonary edema, respiratory failure, or acute non-cardiopulmonary disorder that may affect exercise performance or be aggravated by exercise
* Mental impairment leading to inability to cooperate, provide informed consent, or follow study instructions
* Evidence in the electronic medical record of an absolute contraindication for physical activity
* Severe or advanced orthopedic conditions
* Use of assistive devices for ambulation
* Resides outside of a rural area of Pennsylvania (i.e., one that is not RUCC code 4 - 9 OR RUCA code 4 - 10)
* Pregnant women

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 880 (Estimated)
Dates: Start 2023-05-23 (Actual); Primary Completion 2027-08 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Physical Activity Questionnaire | 12 months vs. baseline
  The 11-question Morgenstern Physical Activity Questionnaire (PAQ-M) is a self-report of physical activity resulting from recreational activities, exercises, home or work activities, and chores.
Objective accelerometry | 12 months vs. baseline
  An accelerometer will be worn for one week to track physical activity.

SECONDARY OUTCOMES:
Physical Activity Questionnaire | 24 months vs. baseline; 24 months vs. 12 months
  The 11-question Morgenstern Physical Activity Questionnaire (PAQ-M) is a self-report of physical activity resulting from recreational activities, exercises, home or work activities, and chores.
Objective accelerometry | 24 months vs. baseline; 24 months vs. 12 months
  An accelerometer will be worn for one week to track physical activity.

CONTACTS AND LOCATIONS:
Overall Officials: Kathryn Schmitz, PhD, Principal Investigator — University of Pittsburgh
Locations (1):
- UPMC, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No